CLINICAL TRIAL: NCT01493167
Title: Study on Circumferential Casting Techniques With WOODCAST
Brief Title: Study on Wood-plastic Composite for Circumferential Casting
Acronym: WOODCAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Onbone Oy (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 37/13/03/02/2011
Record Dates: First submitted 2011-12-13; First posted 2011-12-15 (Estimated); Results first posted 2016-11-15 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2014-12

CONDITIONS: Bone Fracture; Radius Fracture; Ankle Fracture
Keywords: cast; splint; circumferential casting; casting techniques; fracture in extremity
MeSH Terms: conditions — Fractures, Bone; Radius Fractures; Ankle Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- limb casting/splinting (Other): Patient age 0-90 years. Patient treatment requires extremity immobilization
  Interventions: Other: limb casting/splinting

INTERVENTIONS:
Other: limb casting/splinting — ankle and arm cast

SUMMARY:
The purpose of study is to verify that WOODCAST Circular system performs safely and effectively in its intended use.

DETAILED DESCRIPTION:
An ecologically friendly and biodegradable wood-plastic composite-cast is studied. The purpose of the study is to verify that WOODCAST Circular system performs safely and effectively in its intended use. Patients, who need immobilization of extremity (including for example scaphoid fracture of the wrist or ankle fracture) will be participating in the study. Various casting techniques with novel WOODCAST material will be studied.

ELIGIBILITY:
Inclusion Criteria:

* patient treatment involves circular casting;
* age 0-90 years;
* mother tongue finnish or swedish

Exclusion Criteria:

* open fracture;
* other fractures or a previous fracture;
* a previous or simultaneous tendon-, nerve-, or vascular injury to the extremity yo be treated;
* a multiple injured extremity;
* decreased co-operation of the patient;
* malignancy;
* an illness affecting the general health.

Max Age: 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2011-12; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nina C Lindfors, MD PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Limb Casting/Splinting
Started | 97
Completed | 97
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Woodcast Circular System Casts: Operatively treated adult patients needing a post-operative Circular Woodcast scaphoid-type cast
Arm/Group | Woodcast Circular System Casts
Number analyzed (Participants) | 97
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 85
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59
  Male | 38
Region of Enrollment [Number; unit: participants]
  Finland | 97

OUTCOME MEASURES:

1. Primary Outcome: Efficient Casting With Woodcast Circular System
Description: Efficient casting conduc ted with Novel Woodcast material
Time Frame: 1 - 6 weeks
Measure: Number; unit: participants
Arm/Group | Limb Casting/Splinting
Number analyzed (Participants) | 97
participants | 90

ADVERSE EVENTS:
Time Frame: 1-6 weeks (whole treatment period)
Description: All Adverse Events were monitored/collected, but none observed.
Arm/Group | Limb Casting/Splinting
Serious Adverse Events (participants affected / at risk) | 0/97
Other Adverse Events (participants affected / at risk) | 0/97

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No